CLINICAL TRIAL: NCT00842933
Title: An Open-label, Prospective, Randomized, Controlled Clinical Trial of the Use of Reduced Duration Versus Standard Duration Steroid Replacement Therapy for Acute Adrenal Insufficiency in Patients With Septic Shock
Brief Title: Adrenal Insufficiency in Septic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to meet enrollment goal prior to PI transfer
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Laura J Moore, MD, The Methodist Hospital, Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0207-0012
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Septic Shock; Acute Adrenal Insufficiency
Keywords: Septic shock; Acute adrenal insufficiency
MeSH Terms: conditions — Shock, Septic | interventions — Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Corticosteroids discontinued 24 hours after cessation of vasopressor therapy or 7 days, which ever comes first.
  Interventions: Drug: Corticosteroid
- Standard of care group (Active Comparator): Standard corticosteroid therapy given for 7 days as treatment for adrenal insufficiency during septic shock.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — Cessation of corticosteroids 24 hours after cessation of vasopressors
  Other Names: corticosteroids,prednisone,methylpredisolone,hydrocortisone
  Arms: Experimental group
Drug: Corticosteroid — Administer daily for 7 days after diagnosis of acute adrenal insufficiency during septic shock
  Other Names: prednisone,methylprednisolone,corticosteroid,hydrocortisone
  Arms: Standard of care group

SUMMARY:
Randomized controlled trial evaluating the duration of steroid replacement therapy in patients with adrenal insufficiency and septic shock. Patients will be randomized to receive either hydrocortisone 50 mg IV every six hours for seven days (control) or hydrocortisone 50 mg IV every six hours until 24 hours after achievement of hemodynamic stability (MAP > 65 mm Hg off of vasopressors).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older
* Patients who sign informed consent or are represented by a legally authorized representative to provide consent on behalf of the patient
* Patients with septic shock meeting the ACCM/SCCM consensus conference definitions for septic shock

Exclusion Criteria:

* Patients with documented allergic or anaphylactic reactions to corticosteroids
* Patients who have received steroid therapy within 6 months of presentation
* Patients who have received steroids during their hospital admission, with the exception of a single dose of dexamethasone
* Patients who have received etomidate in the preceding 12 hours
* Patients who have had a prior adrenalectomy or a known history of adrenal disease (documented adrenal insufficiency or Cushing syndrome).
* Documented Human Immunodeficiency Virus (HIV) infection
* Pregnancy
* Allergies to adrenocorticotropic hormone (ACTH) or corticosteroids
* Administration of additional medications which may suppress the hypothalamic-pituitary axis:

  * Ketoconazole
  * Aminoglutethimide
  * Mitotane
  * Megestrol acetate
  * Suramin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is the number of hours receiving steroid dosing. | 7 days

SECONDARY OUTCOMES:
A secondary outcome measure will be the difference between daily glucose levels, insulin requirements, and length of stay in the ICU. | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Moore, MD, Principal Investigator — The Methodist Hospital, Houston, TX
Locations (1):
- The Methodist Hospital, Houston, Texas, United States